CLINICAL TRIAL: NCT04865406
Title: Forxiga Tablets General Drug Use-Results Study in Patients With HF
Brief Title: Forxiga HF General Drug Use-Results Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1699C00017
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To capture safety when Forxiga is administered to patients with HF in clinical practice after launch.

DETAILED DESCRIPTION:
The purpose of the study is to review the following points during use of Forxiga Tablets (hereinafter referred to as Forxiga) in the real world setting after launch.

1. ADRs which are unexpected from the precautions for use
2. Understanding of incidence of ADRs during use of Forxiga in the real world setting
3. Factors possibly having an impact on the safety

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 15 years
* Patients who have been prescribed Forxiga for the first time

Exclusion Criteria:

* Patients with a history of hypersensitivity to any ingredients of this drug.
* Patients with severe ketosis, diabetic coma or precoma
* Patients with severe infections, before or after a surgery, or with serious trauma

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic heart failure who use Forxiga for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 1221 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
frequency of adverse drug reactions (ADRs) | 1 year
  Development of ADRs by unexpected from "Precautions for Use" of Forxiga JPI, by SOC, by patient demography and by treatment

CONTACTS AND LOCATIONS:
Locations (45):
- Japan (45):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis Redacted D1699C00017 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1699C00017&attachmentIdentifier=8be28aad-5bbc-486c-9253-ba9ab64bb80e&fileName=CSR_Synopsis_Redacted_D1699C00017.pdf&versionIdentifier=